CLINICAL TRIAL: NCT06221371
Title: Endovascular Treatment With or Without Preceding Intravenous Tenecteplase (TNK) in Patients With Late-window acUte Ischemic Stroke Due to Middle Cerebral Artery Occlusion: a Multi-center, Prospective, Randomized, Open-label, Blinded Endpoint (PROBE), Phase 3 Trial
Brief Title: Endovascular Treatment With or Without Preceding Intravenous Tenecteplase (TNK) in Patients With Late-window acUte Ischemic Stroke Due to Middle Cerebral Artery Occlusion
Acronym: TNK-PLUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Linyi People's Hospital (Other)
Responsible Party: Principal Investigator, Yunyun Xiong, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSA2023YJ003
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Ischemic Stroke, Acute; Thrombolysis; Endovascular Treatment
Keywords: Endovascular Treatment; Thrombolysis; Tenecteplase; Middle cerebral artery occlusion
MeSH Terms: conditions — Ischemic Stroke; Infarction, Middle Cerebral Artery | interventions — Tenecteplase

STUDY DESIGN:
Intervention Model Description: A multi-center, prospective, randomized, open-label, blinded endpoint (PROBE) clinical trial
Who Masked: Outcomes Assessor
Masking Description: blinded-endpoint
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVT with Tenecteplase+EVT (Experimental): Tenecteplase 0.25mg/kg: 1-2 vials (1.0×107 IU/16 mg per vial) Each vial of Tenecteplase is reconstituted with 3 ml sterile water for injection and adjusted to a concentration of 5.33 mg/ml. The total amount of drug will be calculated according to the subject's actual body weight and the required drug volume will be measured. The maximum dose should not exceed 25mg. Tenecteplase should be given as a single, intravenous bolus (drug administered over 5-10 seconds).
  Endovascular treatment (EVT) should be performed as soon as possible after Tenecteplase administration.
  Interventions: Drug: Tenecteplase
- Direct EVT (Active Comparator): During the study period, NMPA-approved stents are permitted. EVT included thrombectomy with stent retrievers, thromboaspiration, intraarterial thrombolysis, balloon angioplasty, stenting, or a combination of these approaches at the discretion of the interventional team.
  Interventions: Device: direct EVT

INTERVENTIONS:
Drug: Tenecteplase — Tenecteplase (0.25 mg/kg, maximum dose 25mg) is given as a single, intravenous bolus (injection over 5 to 10 seconds) immediately upon randomization. EVT should be performed as soon as possible after Tenecteplase administration.
  Arms: IVT with Tenecteplase+EVT
Device: direct EVT — During the study period, NMPA-approved stents are permitted. EVT included thrombectomy with stent retrievers, thromboaspiration, intraarterial thrombolysis, balloon angioplasty, stenting, or a combination of these approaches at the discretion of the interventional team.
  Arms: Direct EVT

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of endovascular treatment with or without preceding intravenous Tenecteplase in patients with late-window (4.5-24 hours of symptom onset) acute ischemic stroke due to middle cerebral artery (MCA) M1 or proximal M2 occlusion.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, patients who meet the inclusion criteria will be randomized to endovascular treatment with preceding intravenous Tenecteplase (0.25mg/kg, maximum 25mg) or without preceding intravenous Tenecteplase in a 1:1 ratio. Written informed consent will be needed.

ELIGIBILITY:
Inclusion criteria

1. Age≥18 years old;
2. Acute ischemic stroke symptom onset between 4.5 to 24 hours prior to enrollment including wake-up stroke and unwitnessed stroke; onset time refers to 'last seen well time';
3. MCA-M1 or proximal M2 occlusions confirmed by Computer Tomography Angiography (CTA)/Magnetic Resonance Angiography (MRA) that was responsible for signs and symptoms of acute ischemic stroke;
4. Neuroimaging: target mismatch profile on CT perfusion (CTP) or MRI + MR perfusion imaging (MRP) (analyzed by perfusion analysis software with Class II and above medical device certificates) [ischemic core volume (defined as CBF<30% or apparent diffusion coefficient value < 620×10-6 mm2/s) <70mL, mismatch ratio≥1.8, mismatch volume≥15mL];
5. Pre-morbid mRS score ≤2;
6. Baseline NIHSS 6-25 (both included);
7. Written informed consent from patients or their legally authorized representative.

Exclusion criteria

1. Patients who decline interventional therapy or intravenous thrombolysis (IVT)；
2. Patients allergic to tenecteplase；
3. Rapidly improving symptoms at the discretion of the investigators；
4. NIHSS consciousness score 1a>2, or epileptic seizure, hemiplegia after seizures or combined with other nervous/mental illness not able to cooperate or unwilling to cooperate；
5. Persistent blood pressure elevation (systolic > 185 mmHg or diastolic >110 mmHg), despite blood pressure lowering treatment；
6. Blood glucose < 2.8 or > 22.2 mmol/L (point of care glucose testing is acceptable)；
7. Active internal bleeding or at high risk of bleeding, e.g.: Major surgery, trauma or gastrointestinal or urinary tract haemorrhage within the previous 21 days, or arterial puncture at a non-compressible site within the previous 7 days；
8. Any known impairment in coagulation, e.g.: If on vitamin K antagonists, then INR >1.7 or prothrombin time >15 seconds; if use of any direct thrombin inhibitors or new oral anticoagulants (NOACs) during the last 48 hours unless reversal of effect can be achieved with idarucizumab; values in sensitivity laboratory tests exceed the upper limit of normal [including activated partial thromboplastin time (APTT), international normalized ratio (INR), platelet count, thrombin time (TT), or appropriate factor Xa activity assays, etc.]; if on heparin during the last 24 hours or with an elevated aPTT greater than the upper limit of normal；
9. Known defect of platelet function or platelet count below 100*109/L (patients on antiplatelet agents can be included)；
10. Ischemic stroke or myocardial infarction in previous 3 months, previous intracranial hemorrhage, severe traumatic brain injury, intracranial or intraspinal operation in previous 3 months, or known intracranial neoplasm (excluding neuroectodermal tumors such as meningioma), arteriovenous malformation or giant aneurysm；
11. Patients who would not be expected to survive more than 1 year；
12. Unable to perform CTP or MRP；
13. Large infarct on non-contrast CT brain or MRI (infarct size >1/3 MCA territory)；
14. Acute or past intracerebral hemorrhage (ICH) identified by CT or MRI, including cerebral parenchymal hemorrhage, intraventricular hemorrhage, subarachnoid haemorrhage, and subdural / extradural hematoma；
15. Multiple arterial occlusions (bilateral MCA occlusion, MCA occlusion accompanied by basilar artery occlusion)；
16. Pregnant women, nursing mothers, or reluctant to take contraceptive measures during the trial period；
17. Unlikely to adhere to the trial protocol or follow-up；
18. Any condition that, in the investigator's judgment, could pose a hazard to the patient if study therapy is initiated or could impact the patient's ability to participate in the study；
19. Participation in any other interventional clinical trials within the previous 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2024-01-25 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2025-10-13 (Actual)

PRIMARY OUTCOMES:
The modified Rankin Scale (mRS) score 0 to 2 at 90 days | 90 days
  The proportion of the modified Rankin Scale (mRS) score 0 to 2 at 90 days. Scores on the mRS range from 0 to 6, with higher scores indicating greater disability.

SECONDARY OUTCOMES:
Ordinal shift analysis of mRS at 90 days (not combined mRS 5 and 6) | 90 days
  Ordinal shift analysis of mRS at 90 days (not combined mRS 5 and 6). Scores on the mRS range from 0 to 6, with higher scores indicating greater disability.
mRS 0-1 at 90 days | 90 days
  The proportion of mRS score 0 - 1 at 90 days. Scores on the mRS range from 0 to 6, with higher scores indicating greater disability.
mRS 0-3 at 90 days | 90 days
  The proportion of mRS 0 - 3 at 90 days. Scores on the mRS range from 0 to 6, with higher scores indicating greater disability.
mRS 5-6 at 90 days | 90 days
  The proportion of mRS 5 - 6 at 90 days. Scores on the mRS range from 0 to 6, with higher scores indicating greater disability.
NIHSS≤1 or a decrease of 8 points or more from baseline at 72h after randomization | 72 hours
  NIHSS≤1 or a decrease of 8 points or more from baseline at 72h after randomization. Scores on the National Institutes of Health Stroke Scale (NIHSS) range from 0 to 42, with higher scores indicating a greater deficit.
Change in stroke severity (NIHSS score) at 7 days after randomization from baseline | 7 days
  Change in stroke severity (NIHSS score) at 7 days after randomization from baseline. Scores on the NIHSS range from 0 to 42, with higher scores indicating a greater deficit.
Successful reperfusion prior to endovascular treatment by DSA (eTICI 2b50-3) | 0 hours (at treatment time)
  Successful reperfusion prior to endovascular treatment by DSA (expanded Treatment in Cerebral Infarction[eTICI] 2b50-3)
Complete recanalization according to CTA or MRA performed 24 hours after randomization | 24 hours
  Complete recanalization according to CTA or MRA performed 24 hours after randomization (arterial occlusive lesion score [AoL]; scale range, 0 [no recanalization] to 3 [complete recanalization]).
Good reperfusion at 24h after randomization | 24 hours
  Good reperfusion at 24h after randomization (Tmax>6s improved by 90% compared with before)

CONTACTS AND LOCATIONS:
Overall Officials: Fengyuan Che, MD, Principal Investigator — Linyi People's Hospital; Yunyun Xiong, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (21):
- China (21):
  - The First Affiliated Hospital of USTC, Hefei, Anhui
  - First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Daxing District People's Hospital, Beijing, Beijing Municipality
  - The 2nd affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Puyang Oilfield General Hospital, Puyang, Henan
  - People's Hospital of Queshan, Zhumadian, Henan
  - First People's Hospital of Chenzhou, Chenzhou, Hunan
  - Dalian Municipal Central Hospital, Dalian, Liaoning
  - First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi
  - Heze Municipal Hospital, Heze, Shandong
  - Jining NO.1 People's Hospital, Jining, Shandong
  - Liaocheng Third People's Hospital, Liaocheng, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Linyi Central Hospital, Linyi, Shandong
  - Qingdao Central Hospital, Qingdao, Shandong
  - Rizhao People's Hospital, Rizhao, Shandong
  - Rizhao Traditional Chinese Medicine Hospital, Rizhao, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Zaozhuang Municipal Hospital, Zaozhuang, Shandong
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang